CLINICAL TRIAL: NCT06488586
Title: In Esketamine and IV Ketamine: Multi-site Observational Study Assessing the Effectiveness and Tolerability of Two Novel Therapies for Treatment-resistant Depression.
Brief Title: IV Ketamine Vs. in Esketamine for MDD TRD
Status: Recruiting | Type: Observational
Sponsor: Gustavo Vazquez (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Envision Mind Care (Unknown); Sunnybrook Health Sciences Centre (Other); Djavad Mowafaghian Centre for Brain Health (Unknown)
Responsible Party: Sponsor-Investigator, Gustavo Vazquez, Professor, Department of Psychiatry, Queen's University, Queen's University
Organization: Queen's University (Other)
Other Study IDs: GHV; Department of Psychiatry. (Other: Queen's University)
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adult outpatients (18-75 years old) with MDD TRD: Participants consisted of adult outpatients (18-75 years old) with unipolar depression experiencing major depressive episodes as determined by the DSM5 and characterized as MDD-TRD, diagnosed with major depressive disorder as outlined by the DSM5 and experienced at least two previous failed antidepressant treatments of adequate dose and duration for the current episode. IV ketamine or IN esketamine are provided as standard-of-care, add-on treatments. Benzodiazepines, naltrexone, lamotrigine, gabapentin and pregabalin, are discontinued prior to the start of the treatment and for the duration of treatment. Patients with psychosis, main diagnosis of personality disorder, uncontrolled hypertension, substance abuse, currently pregnant or breastfeeding, or who had a previous negative reaction to ketamine or esketamine, are ineligible to receive IV ketamine or IN esketamine.
  Interventions: Drug: Low dose IV Ketamine vs. IN Esketamine

INTERVENTIONS:
Drug: Low dose IV Ketamine vs. IN Esketamine — For IV ketamine treatment, ketamine is administered at 0.5mg/kg over 40 minutes. For IN esketamine treatment, esketamine is administered as a nasal spray, two sprays per nostril (56mg total) for the first treatment and three sprays per nostril (84mg) for the rest of the acute series. All treatments are administered at the academic center under the supervision of a mental health care professional. Patients are asked to come fasting at least two hours prior to treatment and to remain resting in the treatment room throughout the dosing session. Throughout each dosing session, blood pressure, oxygen levels, and onset, duration and severity of common side effects are recorded by nursing staff and/or physicians. Patients are discharged after a minimum of 30 minutes post administration, provided that the vital signs return to baseline and that the patient is calm, alert, and oriented.

SUMMARY:
The goal of this observational study is to learn about the comparative acute effects of ketamine vs esketamine in participants over the age of 18 for the treatment of their severe depression and suicidal ideations.

Participants are already taking antidepressants and/or antipsychotics as part of their regular medical care for depression,

DETAILED DESCRIPTION:
This is a multi-center observational prospective cohort study in Providence Care Hospital in Kingston, ON; Envision Mind Care in Edmonton, AB; Center for Addiction and Mental Health in Toronto, ON; the University of British Columbia in Vancouver, BC; and Sunnybrook Health Sciences Center in Toronto, ON, Canada. This study presents real-world clinical data from patients receiving either IV ketamine or IN esketamine for the management of MDD-TRD. Participants consisted of adult outpatients (18-75 years old) with unipolar depression experiencing major depressive episodes as determined by the DSM5 and characterized as MDD-TRD (diagnosed with major depressive disorder as outlined by the DSM5 and experienced at least two previous failed antidepressant treatments of adequate dose and duration for the current episode.

IV ketamine or IN esketamine are provided as standard-of-care, add-on treatments and free of charge to patients. Only medications that have the potential to interact with either ketamine or esketamine, such as benzodiazepines, naltrexone, lamotrigine, gabapentin and pregabalin, are discontinued prior to the start of the treatment and for the duration of treatment. The tapering and discontinuation processes follow the standard-of-care clinical practices and are monitored by the most responsible physician for each patient. Patients with psychosis, main diagnosis of personality disorder, uncontrolled hypertension, substance abuse, currently pregnant or breastfeeding, or who had a previous negative reaction to ketamine or esketamine, are ineligible to receive IV ketamine or IN esketamine.

Approval to perform this study was obtained through the Health Sciences Research Ethics Board at Queen's University (TRAQ #: 6031789). All participants provide voluntary, written informed consent for collecting, analyzing, and presenting aggregate data. This study follows the standards set by the Declaration of Helsinki, and data management complies with US federal Health Insurance Portability and Accountability Act (HIPAA) regulations pertaining to the confidentiality of patient records.

After obtaining informed consent from the participants, Investigators observe participant acute treatment course receiving either IV ketamine or IN esketamine treatment, recording any potential side effects during and after administration and changes in the severity of participant depressive symptoms. In the participating clinical centers, both IV ketamine and IN esketamine treatments consist of bi-weekly sessions for four weeks following standard-of-care clinical guidelines. The decision of delivering IV ketamine or IN esketamine is determined between the patient and the most responsible physician responsible for administering the treatment. Insurance coverage for IN esketamine and patient preference for mode of administration (IV vs IN) are major determinant factors. Since IN esketamine is approved by Health Canada, this is the preferred treatment if a patient has the appropriate insurance coverage, otherwise IV ketamine is offered for free as its cost is covered by the academic center providing the treatment.

For IV ketamine treatment, ketamine is administered at 0.5mg/kg over 40 minutes. For IN esketamine treatment, esketamine is administered as a nasal spray, two sprays per nostril (56mg total) for the first treatment and three sprays per nostril (84mg) for the rest of the acute series. All treatments are administered at the academic center under the supervision of a mental health care professional. Patients are asked to come fasting at least two hours prior to treatment and to remain resting in the treatment room throughout the dosing session. Throughout each dosing session, blood pressure, oxygen levels, and onset, duration and severity of common side effects are recorded by nursing staff and/or physicians. Patients are discharged after a minimum of 30 minutes post administration, provided that the vital signs return to baseline and that the patient is calm, alert, and oriented.

The primary outcome of this study is to determine and compare the clinical effectiveness of IV ketamine and IN esketamine on the management of depressive symptoms using the Montgomery and Åsberg Depression Rating Scale (MADRS). Treatment response is determined as a total score reduction of 50% or more from baseline, partial response to a score reduction between 25% and 50% from baseline score, and remission to a post-treatment MADRS total score of 10 points or less.

Baseline depression symptoms are measured in the week before the first IV ketamine or IN esketamine session. Then progression of depression symptoms through the treatment course is assessed once per week, up to 24 hours after the 2nd, 4th, 6th, and 8th (study endpoint) session. Measurements are performed by an independent trained assessor, not directly involved in the treatment of the patients, virtually or in-person.

The secondary outcome of this study is to determine and compare the effectiveness of IV ketamine and IN esketamine in the reduction of suicidal ideation (SI) and determine the tolerability of these treatments in terms of side effect frequency and severity. The item 10 (Q10) of the MADRS is used to track changes in SI, response is defined as a reduction in Q10 score from baseline to treatment endpoint, and remission as a score of 0 at treatment endpoint (23,25,26). Tolerability of the treatments is regularly assessed during and up to 24 hours after the infusion by the clinic staff and trained independent raters respectively. The assessments include the tracking of depersonalization symptoms using the 6-item Clinician Administered Dissociative Symptom Scale (CADSS-6) (27), dropping out of the treatment, and common side effects associated with these treatments using a checklist: changes in heart rate and blood pressure, anxiety, lightheadedness, drowsiness, dizziness, blurred vision, nausea and headaches. Alterations in the vitals above or below the baseline for each patient are recorded based on severity as mild, medium, or severe following validated clinical guidelines.

Statistical analysis:

The sample size was determined considering the effect size for reduction in depression symptoms for IV ketamine and IN esketamine treatments found in the literature (Cohen's D=1.67 for IV ketamine and Cohen's D=1.24 for IN esketamine), a power of 0.8 and a significance level of p=0.05. Based on these values, Investigators would need a sample size of 24 patients for either treatment to observe a significant effect in a paired sample t-test. The calculations of this study were carried out on IBM SPSS Statistics for Mac, version 24 (IBM Corp., Armonk, N.Y., USA) at a significance level of p<0.05 and applying a per-protocol (only treatment completers) and an intention to treat (ITT) approach for completeness of the analysis and to support the real-world clinical approach of this study. Multiple imputation is applied to address the missing data points, either due to missing assessment questionnaires or patient dropout. The pattern of missing data was random, and Investigators applied a Mersenne Twister algorithm to generate random numbers. This approach conducted 5 multiple imputation iterations using linear regression as the imputation method. Investigators considered the pooled result from the 5 multiple imputation iterations.

For both per-protocol and ITT assessments Investigators analyze the MADRS and CADSS-6 data using descriptive statics and linear regression to compare score changes across different timepoints and between IV ketamine and IN esketamine. For linear regression, Investigators identify the slope and y-intercept coefficient and used correlation coefficient (R2) and P-P plots to determine the goodness of fit of the regression model. Effect size is calculated using Cohen's D (d) with 95% confidence interval (95% CI). Side effect burden is reported in terms of frequency of each side effect and severity (i.e., mild, medium, or severe).

The impact of age and biological sex on treatment response and side effects is analyzed using one-way and two-way multivariate analysis of variance (MANOVA). For this assessment, Investigators assume multivariate normality, homogeneity of covariance matrices, and linearity and employ Wilk's Lambda to test for between-group differences in the multivariate analysis. Post-hoc analysis employs the Tukey's Honest Significant Difference (HSD).

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients (18-75 years old) with unipolar depression experiencing major depressive episodes as determined by the DSM5 and characterized as MDD-TRD (diagnosed with major depressive disorder as outlined by the DSM5) and experienced at least two previous failed antidepressant treatments of adequate dose and duration for the current episode

Exclusion Criteria:

* Individuals with psychosis, main diagnosis of personality disorder, uncontrolled hypertension, substance abuse, currently pregnant or breastfeeding, or who had a previous negative reaction to ketamine or esketamine, were ineligible to receive IV ketamine or IN esketamine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients (18-75 years old) with unipolar depression experiencing major depressive episodes as determined by the DSM5 and characterized as MDD-TRD (diagnosed with major depressive disorder as outlined by the DSM5) and experienced at least two previous failed antidepressant treatments of adequate dose and duration for the current episode
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | From enrollment to the end of treatment at 4 weeks
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which mental health professionals use to measure the severity of depressive episodes in patients with mood disorders.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) item 10 | From enrollment to the end of treatment at 4 weeks
  The Montgomery-Åsberg Depression Rating Scale (MADRS) item 10 is one of the ten-items of this specific questionnaire that assess suicidal thoughts among individuals with depressive episodes (MDD)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo H Vazquez, MD,PhD,FRCPC, Principal Investigator — Queen's University
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gutierrez G, Rosenblat J, Hawken E, Swainson J, Vazquez G. Efficacy and Tolerability of Two Novel "Standard of Care" Treatments-Intranasal Esketamine Versus Intravenous Ketamine-for Treatment-Resistant Depression in Naturalistic Clinical Practice: Protocol for a Pilot Observational Study. JMIR Res Protoc. 2022 May 23;11(5):e34711. doi: 10.2196/34711. PMID 35604752